CLINICAL TRIAL: NCT02011373
Title: Efficacy of IFABONDTM Synthetic Glue for Fixation of Implanted Material in Laparoscopic Sacrocolpopexy: a Prospective Multicenter Study
Acronym: PRO-COLLE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Vitalitec (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013.804
Record Dates: First submitted 2013-12-03; First posted 2013-12-13 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Medial and/or Anterior Genital Prolapse
Keywords: prolapse, laparoscopic sacrocolpopexy, IFABONDTM glue
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IFABOND (Experimental)
  Interventions: Procedure: fixation technique using a sterile synthetic liquid tissue glue: IFABOND™

INTERVENTIONS:
Procedure: fixation technique using a sterile synthetic liquid tissue glue: IFABOND™

SUMMARY:
Laparoscopic sacrocolpopexy is the consensual attitude of choice in genital prolapse but incurs problems of tolerance of implanted material. As an alternative to stapling and suturing, which cause vaginal erosion, we present a fixation technique using a sterile synthetic liquid tissue glue: IFABOND™. A non-randomised prospective multicenter study will assess efficacy in terms of 12-month failure of prolapse correction.

ELIGIBILITY:
Inclusion Criteria:

* Woman aged 18 years or more
* Stage III or IV medial and/or anterior genital prolapse on the Pelvic Organ Prolapse Quantification (POP-Q) classification (hysterocele and/or cystocele), requiring surgical correction
* Patient requesting surgery for the trouble caused by the prolapse

Exclusion Criteria:

* Prolapse of POP-Q stage <III or without functional impact
* Unacceptable postoperative risk disclosed on interview: coagulation disorder, immune disorder, evolutive disease, etc.
* Impaired lower-limb range of motion preventing positioning for surgery
* Pregnancy or intended pregnancy during study period
* Evolutive or latent infection or signs of tissue necrosis on clinical examination
* Non-controlled diabetes (glycated haemoglobin >8%)
* Treatment impacting immune response (immunomodulators), ongoing or within previous month
* History of pelvic region radiation therapy, at any time
* History of pelvic cancer
* Non-controlled evolutive spinal pathology
* Known hypersensitivity to one of the implant components (polypropylene)
* Cyanoacrylate hypersensitivity
* Formaldehyde hypersensitivity
* Inability to understand information provided
* No national health insurance cover; prisoner, or ward of court

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2013-11-06 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Percentage prolapse correction failure | 12 months post-surgery

SECONDARY OUTCOMES:
Percentage prolapse correction failure | 24 months post-surgery
Percentage immediate postoperative failure | 1 month post-surgery
Complications rate | Peroperative and 1, 12 and 24 months post-surgery
Quality of life score | 1, 12 and 24 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Gery Lamblin, MD, Principal Investigator — Gynaecology Department, Hôpital Femme Mère Enfant, Lyon
Locations (3):
- France (3):
  - Gynaecology Department, Hôpital Femme Mère Enfant, Bron
  - Gynaecology Department, Hôpital de la Croix-Rousse, Hospices Civils de Lyon, Lyon
  - Gynaecology Department, Centre Hospitalier Lyon Sud, Hospices Civils de Lyon, Pierre-Bénite

REFERENCES:
- [Result] Lamblin G, Chene G, Warembourg S, Jacquot F, Moret S, Golfier F. Glue mesh fixation in laparoscopic sacrocolpopexy: results at 3 years' follow-up. Int Urogynecol J. 2022 Sep;33(9):2533-2541. doi: 10.1007/s00192-021-04764-4. Epub 2021 Mar 20. PMID 33742249